CLINICAL TRIAL: NCT02712294
Title: Impact of Peripheral Neuromuscular Electrical Stimulation on Spirometry Values, Functional Capacity and Quality of Life in Patients With Pulmonary Hypertension
Brief Title: Impact of NMES on Spirometry Values, Functional Capacity and Quality of Life in Patients With Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Profa. Dra. Vera Lúcia dos Santos Alves, PHD, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Parece 517.472
Record Dates: First submitted 2016-03-08; First posted 2016-03-18 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-02

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; peripheral muscle electrostimulation; capacity of the exercises; quality of life
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (GC) (No Intervention): The GC received standard ambulatory care, including routine exams and drug therapy. All patients were reassessed after the 2 month protocol.
- NMES Group (GE) (Experimental): Receiving the usual care and guidance on their illness, underwent 30 minute NMES sessions twice a week for two months using an electrostimulator. Specifically, 5 cm adhesive surface electrodes in four alternate channels on the Rectus Femoris (two channels the right and two on the left) were used to deliver two-phase symmetrical currents, with a rectangular pulse wave at a frequency of 35 Hz and pulse duration of 250 μ. The time of ascent and descent was one second, contraction time was four seconds and relaxation was eight seconds.
  Interventions: Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation
  Arms: NMES Group (GE)

SUMMARY:
Pulmonary hypertension (PH) features symptoms related to a decreased cardiac autonomic response, pulmonary function and exercise capacity.

Non-pharmacological interventions are low cost and can significant enhance outcomes in these patients. Neuromuscular electrical stimulation (NMES) has been proposed as a viable therapeutic approach in patients with functional limitations, particularly those that present with difficulty to perform exercise protocols.

Objective: to evaluate the impact of NMES on exercise capacity, spirometry values and quality of life of patients with PH.

Material and methods: prospective randomized controlled study with a control group (GC, n9) and NMES goup (GE, n8). Quality of life and exercise capacity through the six-minute walk test (6MWT) were assessed before and after the NMES protocol.

Results: the GE presented with a significant improvement in distance walked in the 6MWT, cycle ergometry, spirometry and quality of life in the areas of vitality, emotional and social aspects of the questionnaire Short Form Health Survey-36.

Conclusion: NMES is a useful tool in the treatment of patients with PH, resulting in improved exercise capacity, quality of life and lung function testing.

ELIGIBILITY:
Inclusion Criteria:

Males and females greater than or equal to 18 years of age, clinically stable with optimized drug therapy in the last 3 months, previously diagnosed with a mean pulmonary arterial pressure ≥ 25 mmHg by right heart catheterization and who agreed to participate by signing an informed consent were included.

Exclusion Criteria:

Exclusion criteria included a diagnosis of Down syndrome, orthopedic disease or neurologic or diagnoses, history of acute heart attack, use of beta-blockers, any urgent or elective surgical intervention during the implementation of the protocol, those who used assistive devices to ambulate or develop an infectious process during the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Distance in six-minute walk test | change from baseline in distance at 2 months
  analysis of distance
Oxygen saturation in six-minute walk test | change from baseline in oxygen saturation at 2 months
  analysis of oxygen saturation at end of test
Systolic blood pressure in six-minute walk test | change from baseline in systolic blood pressure at 2 months
  analysis of systolic blood pressure at end of test
Diastolic blood pressure in six-minute walk test | change from baseline in diastolic blood pressure at 2 months
  analysis of diastolic blood pressure at end of test
Heart rate in six-minute walk test | change from baseline in heart rate at 2 months
  analysis of heart rate at end of test
Borg scale in six-minute walk test | change from baseline in Borg scale at 2 months
  analysis of Borg scale at end of test

SECONDARY OUTCOMES:
The Medical Outcomes Study 36-item Short Form Health Survey | change from baseline at 2 months
  The questionnaire covers 36 items, designed to assess health concepts
Forced vital capacity | change from baseline at 2 months
  spirometric analysis
Forced expiratory volume in the first second | change from baseline at 2 months
  spirometric analysis
Forced expiratory flow 25-75 % | change from baseline at 2 months
  spirometric analysis
Ratio of forced expiratory volume in the first second and forced vital capacity | change from baseline at 2 months
  spirometric analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa of Sao Paulo Medical School, São Paulo, Brazil